CLINICAL TRIAL: NCT02399189
Title: MT-R Followed by Autologous Stem Cells Transplantation in Newly-diagnosed Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Zhu (Other)
Responsible Party: Sponsor-Investigator, Jun Zhu, Chief of the department of lymphoma, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150301
Record Dates: First submitted 2015-03-01; First posted 2015-03-26 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Primary central nervous system lymphoma; rituximab; Methotrexate and Temozolomide; autologous stem cell transplantation; Carmustine and thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-MT followed by auto-HSCT (Experimental): R-MT followed by auto-HSCT Rituximab 375 mg/m2 d1 MTX 3.5g/m2 d2(0.5g/m2 15min,3g/m2 3h） TMZ 100 mg/m2 d2-6 Q21d*4cycles
  Auto-HSCT conditioning regimen:
  BCNU 400mg/m2 d1; Thiotepa 5mg/kg q12h，d2-3
  Interventions: Drug: R-MT followed by auto-HSCT

INTERVENTIONS:
Drug: R-MT followed by auto-HSCT — Four cycles of Induction therapy: Rituximab 375mg/m2 d1; Methotrexate 3.5g/m2 d2;Temozolomide 100mg/m2 d2-6; for patients who reach a CR, PR, or SD, will proceed to autologous stem cell transplantation: Carmustine 400mg/m2 d1; Thiotepa 5mg/kg q12h, d2-3.
  Other Names: Methotrexate(M); Temozolomide(T); Rituximab(R)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of chemotherapy with MT-R followed by autologous stem cells transplantation in newly-diagnosed primary central nervous system lymphoma.

DETAILED DESCRIPTION:
It's a single center, single arm, prospective clinical trial. Patients younger than 65 years old with primary central nervous system lymphoma will received four cycles of chemotherapy with rituximab plus high-dose methotrexate and temozolomide as induction therapy, and then received consolidation therapy with autologous stem cell transplant for which the conditioning regimen is Carmustine plus thiotepa.

ELIGIBILITY:
Inclusion Criteria:

* primary central nervous system diffuse large B-cell lymphoma histologically confirmed by brain biopsy
* ECOG 0-2
* Absence of systemic disease as evaluated by chest-abdomen-pelvis CT scan
* Leucocytes>3.500/mm3, platelets>130.000/mm3, Bilirubin < 2 mg, transaminases < 2.5 N), creatinine < 150 μM/l, creatinine clearance > 50 ml/min/1.73m2
* Age 18-65 years
* Negative HIV test
* Signature of informed consent

Exclusion Criteria:

* prior chemotherapy for primary central nervous system lymphoma
* presence of another cancer (excepting basal cell carcinoma of the skin and cervical carcinoma in situ )
* systemic lymphoma (outside the CNS)
* Isolated ocular lymphoma
* Immunosuppressed patients (HIV , use of immunosuppressors)
* Other uncontrolled or progressive disease compromising shot-term survival
* Severe renal or hepatic disease
* Patients not legally covered by the French Social Security
* Inability to swallow the medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years

SECONDARY OUTCOMES:
overall response rate | 2 years
overall survival | 2 years
event-free survival | 2 years

OTHER OUTCOMES:
neurotoxicity | 2 years
  using a battery of cognitive and quality-of-life (QoL) measures

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Lijuan Deng, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Correa DD, Maron L, Harder H, Klein M, Armstrong CL, Calabrese P, Bromberg JE, Abrey LE, Batchelor TT, Schiff D. Cognitive functions in primary central nervous system lymphoma: literature review and assessment guidelines. Ann Oncol. 2007 Jul;18(7):1145-51. doi: 10.1093/annonc/mdl464. Epub 2007 Feb 6. PMID 17284616